CLINICAL TRIAL: NCT04701502
Title: Efficacy and Safety of Viusid and Asbrip in Hospitalized Patients With Mild and Moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: COVID_BULG_2020
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Respiratory Disease; Immune System; Immunomodulator; Antiseptic; Supportive Care
MeSH Terms: conditions — COVID-19; Respiration Disorders | interventions — Viusid; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): A total of 60 subjects will be randomized 2: 1 in this study. 40 patients will be assigned to Viusid plus Asbrip, plus standard care of the hospital.
  Treatment duration: 21 days.
  Interventions: Dietary Supplement: Viusid; Dietary Supplement: Asbrip; Drug: Standard Care
- Control (Other): A total of 60 subjects will be randomized 2: 1 in this study. 20 control patients will be assigned to standard care of the hospital only.
  Treatment duration: 21 days.
  Interventions: Drug: Standard Care

INTERVENTIONS:
Dietary Supplement: Viusid — Patients received daily doses of 30 ml of Viusid every 8 hours plus standard care for COVID-19. Viusid is administered orally.
  Treatment duration: 21 days
  Arms: Interventional
Dietary Supplement: Asbrip — Patients received daily doses of 10 ml of Asbrip every 8 hours plus standard care for COVID-19. Asbrip is administered orally.
  Treatment duration: 21 days
  Arms: Interventional
Drug: Standard Care — Standard care for COVID-19

SUMMARY:
This is a two-arm, randomized, open label, two-center, controlled study to evaluate the safety and efficacy of Viusid plus Asbrip in patients with mild and moderate symptoms of respiratory illness caused by Coronavirus 2019 infection.

DETAILED DESCRIPTION:
This is a two-arm, randomized, open label, two-center, controlled study to evaluate the safety and efficacy of Viusid plus Asbrip in patients with mild and moderate symptoms of respiratory illness caused by Coronavirus 2019 infection.

A total of 60 subjects will be randomized 2:1 in this study. 40 patients will be assigned to receive daily oral doses of 30 ml of Viusid and 10 ml of Asbrip every 8 hours and standard care. Other 20 patients will be assigned to receive only standard care.

Treatment duration: 21 days

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults aged ≥18 years at the time of enrollment.
2. Subjects with mild-to-moderate symptoms of respiratory illness caused by coronavirus 2019 infection as defined below:

   Mild (uncomplicated) Illness:
   * Diagnosed with COVID-19 by a standardized RT-PCR assay and
   * Mild symptoms, such as fever, rhinorrhea, mild cough, sore throat, malaise, headache, muscle pain, or malaise, but with no shortness of breath and
   * No signs of a more serious lower airway disease and
   * RR<20, HR <90, oxygen saturation (pulse oximetry) > 93% on room air

   Moderate Illness:
   * Diagnosed with COVID-19 by a standardized RT-PCR assay and
   * In addition to symptoms above, more significant lower respiratory symptoms, including shortness of breath (at rest or with exertion) or
   * Signs of moderate pneumonia, including RR ≥ 20 but <30, HR ≥ 90 but less than 125, oxygen saturation (pulse oximetry) > 93% on room air and
   * If available, lung infiltrates based on X-ray or CT scan < 50% present
3. Clinically normal resting 12-lead ECG at screening visit or, if abnormal, considered not clinically significant by the Principal Investigator.
4. Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.
5. Understands and agrees to comply with planned study procedures.

Exclusion Criteria:

1. Subjects showing signs of acute respiratory distress syndrome (ARDS) or respiratory failure necessitating mechanical ventilation at the time of screening.
2. History of severe chronic respiratory disease and requirement for long-term oxygen therapy.
3. Subjects showing signs of clinical jaundice at the time of screening.
4. History of moderate and severe liver disease (Child-Pugh score >12).
5. Subjects requiring Renal Replacement Therapy (RRT) at the time of screening.
6. History of uncontrolled diabetes.
7. History of severe chronic kidney disease or requiring dialysis.
8. Any uncontrolled active systemic infection requiring admission to an intensive care unit (ICU); Note: Subjects infected with chronic hepatitis B virus or hepatitis C virus will be eligible for the study if they have no signs of hepatic decompensation.
9. Patients with malignant tumor, or other serious systemic diseases.
10. Patients who are participating in other clinical trials.
11. Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Viusid or Asbrip are not eligible.

Note: Empirical antibiotic treatment for secondary bacterial infections is allowed during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Clinical Improvement | 21 days
  Clinical Improvement as assessed by change in total symptom score ranging from 0-12.
  The symptom score includes: [everyday assessment, up to 21 days].
  1. Fever (temperature in oC) based on a scale 0-3: 0 <36,7; 1 =36,7-37,8; 2 =37,8-38,9; 3 > 38,9.
  2. Cough on a scale 0-3: 0 = no cough, 1 = mild, 2 = moderate, 3 = severe.
  3. Shortness of breath based on a scale 0-3: 0 = no shortness of breath, 1 = with moderate intensity exercise, 2 = with walking on flat surface, 3 = short of breath with getting dressed or daily activities.
  4. Fatigue on a 0-3 scale: 0 = no fatigue, 1 = mild fatigue, 2 = moderate fatigue, 3 = severe fatigue.
  Composite score is a sum of mentioned four symptom scores, assessed every day up to 21 days. It ranges from 0 to 12.
Time to semirecover | 21 days
  Efficacy will be determined by the number of days required to reach a 50 percent reduction in the composite score, i.e. "time to semirecovery" (primary outcome measure).
Symptom resolution | 21 days
  Symptom resolution of COVID-19 disease The number of days required to reach symptom score <0,25 for each one of four symptom category mentioned before.
Time to recovery | 21 days
  Time (days) to recovery from COVID-19 disease The number of days required to reach composite score <1.

SECONDARY OUTCOMES:
Cumulative assessment of disease severity | 21 days
  Disease severity will be measured using a disease severity clinical event scale (assessed until day 21) Change from baseline in the patient's health status on an ordinal scale of 7 categories.
  1. Death
  2. Hospitalized, with invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, with non-invasive ventilation or high-flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, which does not require supplemental oxygen
  6. Not hospitalized, limitation of activities.
  7. Not hospitalized, without limitations in activities. Note: lower scores mean a worse result.
  Note: lower scores mean a worse outcome
Duration of SARS-CoV-2 PCR positivity | 21 days
  Daily PCR analysis to measure and compare viral load
Concentration of C-reactive protein in peripheral blood | 21 days
  Concentration of C-reactive protein in peripheral blood measured by Blood biochemical analysis.
Incidence of hospitalization | 21 days
  Number of Incidence of hospitalization
Duration (days) of hospitalization | 21 days
  Number of days of hospitalization
Incidence of mechanical ventilation supply | 21 days
  Number of incidences of mechanical ventilation supply per patient
Incidence of oxygen use | 21 days
  Number of incidences of oxygen use
Duration (days) of oxygen use | 21 days
  Number of days of oxygen use per patient
Mortality rate | 21 days
  Number of death per group

OTHER OUTCOMES:
Change in liver function test | 21 days
  Change in liver function test (AST, ALT and TBIL) by blood biochemical analysis.
Change in kidney function test | 21 days
  Change in kidney function with creatine clearance rate by blood and urinary biochemical analysis.
Change in routine blood test | 21 days
  Change in routine blood test red blood cells concentration by blood biochemical analysis.
Change in routine blood test | 21 days
  Change in routine blood test white blood cell concentration by blood biochemical analysis.
Change in routine blood test | 21 days
  Change in routine blood test D-dimer level by blood biochemical analysis.
Change in routine blood test | 21 days
  Change in routine blood test fibrinogen level by blood biochemical analysis at day.

CONTACTS AND LOCATIONS:
Locations (2):
- Bulgaria (2):
  - MBAL, Sv. Mina, Plovdiv
  - MTB Plovdiv, Plovdiv

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR